CLINICAL TRIAL: NCT03805477
Title: Nintedanib in Patients With Bronchiolitis Obliterans Syndrome Following Hematopoietic Stem Cell Transplantation (HSCT)- a Multicentre Phase II Trial
Brief Title: Nintedanib in Patients With Bronchiolitis Obliterans Syndrome Following Hematopoietic Stem Cell Transplantation
Acronym: NINBOST2018
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00837; me17Hostettler
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bronchiolitis Obliterans Syndrome (BOS); Bronchiolitis Obliterans (BO)
Keywords: allogeneic hematopoietic cell transplantation.; chronic graft-versus-host disease (cGvHD); Nintedanib; fibrotic lung disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nintedanib (Experimental): Nintedanib 150 mg Kps bid (oral)
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib 150 mg Kps bid (oral); in order to manage adverse events, the dose of Nintedanib may be reduced from 150 mg twice daily to 100 mg twice daily

SUMMARY:
This study investigates the safety and tolerability of Nintedanib in patients with bronchiolitis obliterans syndrome (BOS) following allogeneic hematopoietic cell transplantation. All study patients with BOS will be treated with the study drug Nintedanib (300 mg/day) as an add-on therapy to their basic immunosuppressive treatment over a 12-months treatment period.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HCT) is an established treatment option for several malignant and non-malignant disorders. An important limitation of long-term survival after HCT is chronic graft-versus-host disease (cGvHD). The manifestation of cGvHD in the lungs, bronchiolitis obliterans (BO - if proven by lung biopsy) or bronchiolitis obliterans syndrome (BOS - clinical diagnosis), has a reported incidence between 5 and 20%. Despite different treatment approaches, prognosis of BO remains poor, with an overall 3-year mortality of up to 65%. Nintedanib is an orally available indolinone derivate that competitively binds to the vascular endothelial growth factor (VEGF) receptors, fibroblast growth factor (FGF) receptors, and platelet derived growth factor (PDGF) receptors. The anti-fibrotic activities of Nintedanib may impact the progressive course of fibrotic lung diseases like BO. This study investigates the safety and tolerability of Nintedanib in patients with bronchiolitis obliterans syndrome following allogeneic hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Time interval from transplant </= 5 years at the time of inclusion
* BOS as defined per the National Institute of Health (NIH) criteria:

  1. FEV1/vital capacity < 0.7 or the fifth percentile of predicted.
  2. FEV1 < 75% of predicted with ≥ 10% decline over less than 2 years.
  3. Absence of infection in the respiratory tract, documented with investigations directed by clinical symptoms, such as chest radiographs, computed tomographic (CT) scans, or microbiologic cultures (sinus aspiration, upper respiratory tract viral screen, sputum culture, and broncho-alveolar lavage).
  4. One of the 2 supporting features of BOS: 1. Evidence of air trapping by expiratory CT or small airway thickening or bronchiectasis by high-resolution chest CT, or 2. Evidence of air trapping by PFTs: residual volume > 120% of predicted or residual volume/total lung capacity elevated outside the 90% confidence interval and prior or current diagnosis of cGvHD per NIH criteria or histologically proven BO
* Diagnosis of BOS within 6 months before enrollment or prior diagnosis of BOS with an absolute decline of the percentage of predicted forced expiratory volume in 1 second (FEV1) by >/= 10% within the past 12 months before inclusion

Exclusion Criteria

* Known intolerance to Nintedanib or any of its component
* Pregnancy or nursing
* Serum ALT > 5 x upper limit of normal (ULN) unless explained entirely by liver GvHD or total bilirubin > 3x ULN unless explained entirely by liver GvHD
* Any acute pulmonary infection with viruses, bacteria or fungi within four weeks before study inclusion
* Chronic oxygen therapy; non-invasive ventilation
* Inability to give informed consent or to perform repeated pulmonary function tests (PFT)
* Life expectancy < 1 year at the time of enrolment as suggested by the treating physician
* Hematologic malignancy in hematologic relapse
* Symptomatic angina pectoris
* Therapeutic anticoagulation (primary or secondary prophylactic platelet anti-aggregation allowed)
* Recent abdominal surgery or untreated gastric ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
adverse event rate leading to interruption/ discontinuation of study treatment | from screening to month 12 after screening
  adverse events of the following severity according to Common terminology criteria for adverse events(CTCAE): Diarrhoea ≥ grade 3; Nausea ≥ grade 3; Vomiting ≥ grade 3; Abdominal pain ≥ grade 3; Elevation of liver enzymes (AST, ALT) ≥ grade 2; Elevation of total bilirubin ≥ 2

SECONDARY OUTCOMES:
change of the percent of predicted forced expiratory volume in 1 second (FEV1) | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  absolute change of the percent of predicted FEV1 by ≥10% from FEV1 before enrolment (eg, 50% to 40% predicted FEV1), confirmed by 2 pulmonary function tests (PFT) performed at least two weeks apart and after exclusion of infections and extra pulmonary causes
change in forced vital capacity (FVC) | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  volume of air that can forcibly be blown out after full inspiration, (measured in Liters)
change in total lung capacity (TLC) | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  the volume in the lungs at maximal Inflation (measured in liters)
Change in diffusion capacity of the lung for carbon monoxide (DLCO) | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  extent to which oxygen passes from the air sacs of the lungs into the blood (measured in "ml/min/kPa)
Change in exhaled nitric oxide (eNO) | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  Change in exhaled nitric oxide (eNO) (measured in parts per Billion)
Nitrogen (N2)-washout | Pulmonary function tests will be performed at screening, after 1, 2, 3, 6, 9, 12 and after 13 months
  The following describes a single-breath nitrogen test: A subject takes a breath of 100% oxygen and exhales through a one-way valve measuring nitrogen content and volume. A plot of the nitrogen concentration (as a % of total gas) vs. expired volume is obtained by increasing the nitrogen concentration from zero to the percentage of nitrogen in the alveoli. The nitrogen concentration is initially zero because the subject is exhaling the dead space oxygen they just breathed in (does not participate in alveolar exchange), and climbs as alveolar air mixes with the dead space air. The dead space can be determined from this curve by drawing a vertical line down the curve such that the areas below the curve (left of the line) and above the curve (right of the line) are equal
changes in in 6 minutes walking distance (6-MWD) | 6-MWD will be performed at screening, after 6, after 12 months
  standardized 6-minute walk test will be performed breathing room air and performed according to the guidelines of the American Thoracic Society. Significant drop of transcutaneous measured arterial oxygen Saturation (SaO2) is defined as a ΔSaO2 ≥ 4% or SaO2 < 90%. A significant change in walking distance will be Δ distance = 40 metre.
cumulative steroid doses | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  steroid doses per month (in mg)
occurrence of GvHD in other organs | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  occurrence of GvHD in other organs
disease-free survival of underlying hematologic disease | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  disease-free survival of underlying hematologic disease
changes in St. George's Respiratory Questionnaire (SGRQ) | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  The SGRQ is designed to measure health impairment in patients with asthma and chronic obstructive pulmonary disease (COPD); 3 component scores are calculated: symptoms; activity; impacts. Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100.
changes in NIH GvHD grading score | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  NIH symptom-based lung score (score 0: no symptoms, score 1: shortness of breath with stairs, score 2: shortness of breath on flat ground, score 3: shortness of breath at rest or requiring oxygen)
changes in Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) questionnaire | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  specific HSCT-patients validated self-report questionnaire using a 5 point Likert scale and covering 4 specific domains that include physical, social and family, emotional and functional well-being. Scoring produces a range from 0-148, the higher the score, the better the Quality of Life (QOL).
overall survival | assessed at screening, after 1, 2, 3, 6, 9, 12, and after 13 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Hostettler Haack, PD Dr. med, Principal Investigator — Clinic of Respiratory Medicine, University Hospital Basel
Locations (3):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Switzerland (2):
  - Clinic of Hematology, University Hospital Basel, Basel
  - Clinic of Respiratory Medicine, University Hospital Basel, Basel